CLINICAL TRIAL: NCT06066255
Title: REINFORCED PROPHYLAXIS OF GVH IN ELDERLY PATIENTS WITH HAEMATOLOGICAL MALIGNANCIES RECEIVING HAPLOIDENTICAL ALLOGENEIC HEMATOPOIETIC STEM CELL TRANSPLANTATION: USE OF A LOW DOSE OF POST-ALLOGRAFT ANTI-LYMPHOCYTIC SERUM
Brief Title: PROPHYLAXIS OF GVH IN ELDERLY PATIENTS RECEIVING HAPLOIDENTICAL ALLOGENIC HEMATOPOIETIC STEM CELL TRASNPLANTATION USE OF A LOW DOSE ANTI-LYMPHOCYTIC SERUM
Acronym: CASPER
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CASPER-ATG-IPC 2023-015
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hematological Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Thymoglobulin Injectable Product — single intravenous injection of thymoglobulin

SUMMARY:
The aim of this trial is to evaluate the efficacy of GVH prophylaxis reinforced by low-dose Thymoglobulin administered at the end of aplasia after haploidentical allogeneic transplantation.

Patients will receive a single infusion of Thymoglobulin at a dose of 1 mg/kg between 48h and 72h after emergence from aplasia, and will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 60 or aged 50 to 59 with comorbidities (HCT-CI10 score ≥ 3),
* Hematological malignancies except myeloproliferative syndrome and myelodysplastic syndrome,
* Patient having received an allograft within ≤ 35 days, performed with the following modalities:

  * First allogeneic transplant,
  * Haploidentical donor,
  * Peripheral stem cell transplant,
  * Non-myeloablative "Baltimore"-type conditioning, delivered as standard in routine care, as reported in the literature (fludarabine, cyclophosphamide, total body irradiation),
  * Standard GVHD prophylaxis in the context of haploidentical transplants (post-transplant cyclophosphamide, ciclosporin A and mycophenolate mofetil).
* Patient discharged from aplasia within ≤ 35 days,
* Signed informed consent form,
* Affiliation with a social security.

Exclusion Criteria:

* Previous allogeneic or organ transplant,
* Presence of signs of GVHD,
* Contraindications to treatment with Thymoglobuline®,
* Hypersensitivity to rabbit proteins or to any of the excipients listed in the "Composition" section of the summary of product characteristics,
* Pregnant women or may become pregnant (without effective contraception) or breast-feeding,
* Persons in emergency situations or unable to give informed consent form,
* Adult with a legal protection measure (adult under guardianship, curatorship or safeguard of justice),
* Unable to comply with medical follow-up for geographical, social or psychological reasons.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-03-31 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of acute GVH | Day 100
  To assess the rate of grade 2-4 acute GVHD post allograft using the MAGIC classification.

SECONDARY OUTCOMES:
Acute GVH | day(D) 30, D60, D90, D100, D120, D180, D270 and D365
  Grade 2-4 acute GVHD will be assessed using the MAGIC classification post allograft
chronic GVH | day(D)100, D120, D180, D270 and D365
  Chronic GVHD will be assessed using NIH classification post allograft,
Cumulative incidence of chronic GVH | 1 year
  Cumulative incidence of chronic GVHD at 1 year post-transplant,
Cumulative incidence of NRM | 1 year
  Cumulative incidence of NRM at 1 year post-transplant,
Cumulative incidence of relapse | 1 year
  Cumulative incidence of relapse at 1 year post-transplant,
Immunology | day(D)100, D120, D180, D270 and D365
  Blood T, B and NK lymphocyte counts post-transplant,
Viral infections | between day (D)30 and D120
  Cumulative incidence of invasive fungal and viral infections (CMV, EBV, BK virus) post allograft,
Cumulative incidence | Day 100
  Cumulative incidence of EBMT-defined "poor graft function" post-transplant.
Survival | 1 year
  Progression-free survival and overall survival at 1 year post-transplant,

IPD SHARING:
Plan to Share IPD: No